CLINICAL TRIAL: NCT03252444
Title: Therapeutic Approaches for Subjects With Scapula Dyskinesis: Conscious Control, EMG Biofeedback Training, and Intensive Scapula-focused Intervention
Brief Title: Therapeutic Approaches for Subjects With Scapula Dyskinesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201412043RINA
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2017-08

CONDITIONS: Shoulder Impingement
Keywords: Shoulder dyskinesis; EMG biofeedback training; Intensive Scapula-focused intervention
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback group (Experimental): After 1 minute of rest, participants will perform 6 trials of bilateral, active, weighted arm elevation in the scapular plane and a therapist classifies the scapular motion into specific patterns of scapular dyskinesis. After the evaluation of scapular dyskinesis, the kinematics and surface EMG (sEMG) data will be collected during 5 trials of the same arm movements and 3 selected exercises.
  Interventions: Other: Conscious control+biofeedback
- Conscious control group (Active Comparator): Conscious correction of scapular orientation will be taught to the subjects in the manner described in previous studies. The starting position is determined in each individual by actively positioning the scapula between maximal upward and downward rotation, external and internal rotation, and posterior and anterior tilt. Scapular assistance test (SAT) is also conducted by passively assisting patients' scapula into appropriate position to correct scapula dyskinesis
  Interventions: Other: Conscious control

INTERVENTIONS:
Other: Conscious control — Conscious control of the scapula is important and can correct neuromuscular coordination as well as strength deficits. The strategy in learning control of scapula into normal orientation can be facilitated by manual guides and/or external cues
  Arms: Conscious control group
Other: Conscious control+biofeedback — In electromyography (EMG) biofeedback training, electronic equipment is used to reveal instantaneously certain physiological events.
  Arms: Biofeedback group

SUMMARY:
The investigators will test whether conscious control with manual guides and video or EMG biofeedback will enhance 3-D kinematics of scapula in shoulder dysfunction subjects with different type of scapula dyskinesis. The investigators will also examine how correction of scapular orientation may affect the activation of associated muscles during various dynamic movements in these subjects.

ELIGIBILITY:
Inclusion criteria:

* At least three positive of five tests, including Neer's test, Hawkin's test, Empty can test, tenderness in tendon of rotator cuff and resisted external test.
* Each patient will need a prescription of the physician or orthopedic surgeon for diagnosing impingement symptoms

Exclusion criteria:

- Shoulder pain onset due to trauma, a history of shoulder fractures or dislocation, cervical radiculopathy, degenerative joint disease of the shoulder, surgical interventions on the shoulder, or inflammatory arthropathy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2017-05-21 (Actual); Study Completion 2017-05-21 (Actual)

PRIMARY OUTCOMES:
Shoulder complex kinematics | The scapular kinematics will be measured before scapular control and immediately after scapular control
  Scapular orientation relative to the thorax is described using a Euler angle sequence of rotation about Zs (protraction/retraction), rotation about Y's (downward /upward rotation), and rotation about X"s (posterior/anterior tipping). Scapular elevation is defined as the vertical displacement of the scapular sensor during arm elevation. Humeral orientation relative to the scapula is described using a Euler angle sequence in which the first rotation represents the plane of elevation, the second rotation defines the amount of elevation, and the third rotation describes the amount of axial rotation.
Shoulder associated muscular activities | The muscle activation will be measured before scapular control and immediately after scapular control
  Full bandwidth sEMG data, captured by data acquisition software (AcqKnowledge, Biopac systems Inc., CA, USA)

SECONDARY OUTCOMES:
Forward shoulder posture | After subjects are included in the study, the forward shoulder posture will be measured before scapular control, and be done within 2 hours.
  The measurement of the distance between the posterior border of the acromion and the table
Pectoralis minor muscle length | After subjects are included in the study, the muscle length will be measured before scapular control, and be done within 2 hours.
  The distance from the fourth rib to the coracoids process will be measured with FASTRAK system with accuracy of 0.08 cm. This distance (in centimeter) is divided by the subjects height and multiplied by 100. This results in a pectoralis muscle length index

CONTACTS AND LOCATIONS:
Overall Officials: Jiu- Jenq Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Du WY, Huang TS, Chiu YC, Mao SJ, Hung LW, Liu MF, Yang JL, Lin JJ. Single-Session Video and Electromyography Feedback in Overhead Athletes With Scapular Dyskinesis and Impingement Syndrome. J Athl Train. 2020 Mar;55(3):265-273. doi: 10.4085/1062-6050-490-18. Epub 2019 Dec 26. PMID 31876455